CLINICAL TRIAL: NCT04851704
Title: Child Self-regulation: Impact and Neurocognitive Underpinnings of a Psychosocial Intervention
Brief Title: Child Self-regulation: A Pilot Study on the Impact of Tuning in to Kids Parent Intervention
Acronym: N-TIK Pilot
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Evalill Bølstad, PhD, Associate Professor, University of Oslo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015/2383 REK
Record Dates: First submitted 2021-04-14; First posted 2021-04-20 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Parent and Child Emotional Intelligence and Child Self-regulation
Keywords: Tuning in to Kids; Parent Interventions; Child self-regulation

STUDY DESIGN:
Intervention Model Description: Intervention-control trial, where both intervention and control group participants are assessed at baseline, and then the intervention groups get the intervention, and all group participants are assessed at follow up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Tuning in to Kids parenting program (Experimental): Intervention groups receive the Tuning in to Kids parenting program
  Interventions: Behavioral: Tuning in to Kids
- Control: Business as usual (No Intervention): Control groups have "business as usual", and then get offered the intervention program after 6 months follow-up assessment.

INTERVENTIONS:
Behavioral: Tuning in to Kids — A parenting program that includes 6 group supervisions of parents, where emotion coaching and promotion of kids emotional competence are main focus.
  Arms: Intervention: Tuning in to Kids parenting program

SUMMARY:
The current pilot project will a) adapt an evidence-based psychosocial intervention program and conduct a randomized controlled trial with a group of Norwegian parents of preschool children, b) evaluate the intervention'simpact on child mental health and c) investigate the cognitive and physiological underpinnings of this effect.This pilot study will recruit 40 Norwegian parents of preschool children prior to the transition to starting school. Baseline measures will include parent emotion coaching and parent functioning, child emotion regulation, social and behavioral functioning, child behavioral and physiological indices of cognitive capacity and attention functioning, and school adjustment. Following completion of baseline assessment, parents will be randomized into Intervention or Wait-list conditions. Intervention parents will attend a 6-session group parenting program where they will learn to emotion coach their children and regulate their own emotions. Post-program, Intervention parents will complete program evaluation to determine program feasibility and acceptability. At 6-month follow-up baseline assessments will be repeated for Intervention and Wait-list participants with primary school teachers reporting on children's adjustment to school. Wait-list parents will then be offered the N-TIK program.

DETAILED DESCRIPTION:
Promoting the emotional functioning of preschool children prior to the transition to school has important implications for their adjustment and mental health. Parents can assist children to understand and regulate their emotions thereby better equipping the child as they face this often highly stressful and anxiety provoking period. In addition, we need more knowledge on how processes on both behavioral and physiological levels can contribute to explain the mechanisms underlying changes in child self-regulation influenced by parents and the home environment.

Thus, a 2 x 2 intervention design pilot study of the Norwegian version of Tuning in to Kids (N-TIK) comparing intervention and wait-list participants will examine:

i) Does N-TIK lead to better parent-reported parent emotion coaching? ii) Does N-TIK lead to better parent-reported child emotional competencies, mental health and adjustment? iii) Does N-TIK lead to improved child attentional and executive functions as measured by behavioral performance and changes in neural and pupillometric responses in experimental tasks? The intervention aims to improve the responsiveness of parents to emotions, both in themselves and their children. Theoretically, this is anticipated to lead to children developing greater awareness and knowledge of their own emotional experience, to reduced levels of emotionality, and to greater internal self-awareness of their emotions (cognitive awareness about emotional experience). These comprise some of the core emotional competencies relevant for enhancing the transition to school. In turn these competencies are anticipated to be related to greater emotional, cognitive and physiological regulation as assessed by experimental paradigms and physiological measures. For children at risk (due to limited emotional, cognitive, physiological and behavioural regulation), an intervention that assists their parents to learn specific skills that enhance their emotion-related parenting, these risks are likely to be mitigated.

This study will be highly innovative on several counts. It will: gather preliminary evidence using a 2 x 2 intervention design for the effectiveness of an emotion-focused parenting program using a Norwegian sample; use cutting-edge behavioral and physiological measures to see whether participation in N-TIK leads to improved child attentional and executive functions - critical skills that assist with learning and self-regulation; integrate important disciplines within psychology by combining an intervention including preventive actions with emotional, neurocognitive and physiological approaches within adevelopmental psychological framework.

Statistical Analyses Time 1 data will be examined to determine relationships between key constructs. ANCOVA will be used to examine changes over time and to compare Intervention and Wait-list participants on all outcomes.

Ethical aspects The research will be carried out according to the Helsinki declaration, and we will go to great lengths to ensure proper ethical treatment. The potential risks involved in this study relate to where concerns might arise with parents, or where parents have specific difficulties with children: 1. Families who show significant levels of distress and difficulty during the program will have access to appropriate support and intervention services. If during the research period the investigators believe that either the children or the parents are experiencing serious psychological difficulties, if issues of abuse are suspected, or if parents themselves request support or intervention, the investigators will discuss with the family what appropriate professional intervention services are available, and assist in a referral. 2. Issues of confidentiality: Because many of the sample will be recruited from preschool classes, teachers and other parents will be aware of individuals who are part of the research and the groups. Teachers will not be given information gained from the parents. At the beginning of each of the six sessions, parents will be reminded that all material or issues discussed in groups remains confidential and should not be discussed with anyone outside of the group. Issues of confidentiality will only be broken should the research investigators feel that either a child or parent is at undue risk of being harmed/or harming others. Should this occur, parents and children will be fully informed about the processes involved in initiating assistance. 3. The specific methods used in this research are unlikely to be a potential risk to participants. The questionnaires used in the assessment have been widely used in previous research, and have been found not to cause undue concern. The home observation task requires the parent and child to read a story together and talk about the emotions in the story while being videotaped. This is not thought to be likely to cause undue concern. However, if parents find any material in the group, questionnaires, or home observation causes them any difficulty, they will be encouraged to talk with one of the two group leaders and/or to contact the research investigators, and they will be offered referrals to appropriate services should these be required. There are no risks associated with the laboratory assessment.4. The research involves a wait-list control group where half the participants are assigned to wait for a six-month period before receiving the intervention. Should any problems occur during this six-month period, the study investigators would refer the family for appropriate assistance. 5. Should any of the material or exercises performed in the group cause undue concern, immediate debriefing with the group leaders will be provided.

The applicant, Dr Karevold, is an authorized clinical psychologist and thus legally obliged to follow the Health Personnel Act. All research activities will be performed accordingly to ensure participants' personal integrity and health. General guidelines for research will be followed.

ELIGIBILITY:
Inclusion Criteria:

* A preschool child aged 5-6 years old
* Parent of a preschool child aged 5-6 years old

Exclusion Criteria:

* Parents under the age of 18
* Parents not able to read and write in Norwegian

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Parent Emotional Style Questionnaire (PESQ) | Six months: Change in PESQ from baseline to follow up 6 months after baseline measured by questionnaire reports.
  Parent Emotion Socialization Questionnaire (PESQ) is a scale with items that are scored from 1 to 5, where 5 indicates high levels of specific parenting beliefs (i.e. emotion coaching and emotion dismissive beliefs).
Coping with children negative emotions scale (CCNES) | Six months: Change in CCNES from baseline to 6 months follow-up measured by questionnaire reports.
  Coping with children negative emotions scale (CCNES) is a scale with items that are scored from 1 to 7, where 7 indicates high levels of specific parenting behavior (i.e. supportive and nonsupportive parenting behavior).
Eysenck's child behavior questionnaire (ECBI) | Six months: Change in ECBI from baseline to 6 months follow-up measured by questionnaire reports.
  Eysenck's child behavior questionnaire (ECBI) is a scale with items that are scored from 1 to 7, where 7 indicates high levels of behavior problems.
Preschool anxiety scale - revised (PAS-R) | Six months: Change in PAS-R from baseline to 6 months follow-up measured by questionnaire reports.
  Preschool anxiety scale - revised (PAS-R) is a scale with items that are scored from 1 to 5, where higher score indicates higher levels of anxiety.
Emotional Go/Nogo task (EGNG) | Six months: Change in EGNG from baseline to 6 months follow-up measured by lab assessment.
  EGNG is a direct assessment of child behavior - an adaptation from the Go/NoGo task - a well-established cognitive paradigm. When modified with emotional stimuli in the form of faces with different positive and negative emotional expressions serving as either target or non-target, the task allows for behavioural assessment of emotion discrimination, emotion regulation and cognitive control, which are related, yet separable processes (Tottenham et al. 2011).
AX Continuous Performance Task (AX-CPT) | Six months: Change in AX-CPT from baseline to 6 months follow-up measured by lab assessment.
  AX-CPT is a direct assessment of child behavior - The AX-CPT task (a version of the classic Continuous Performance Test, Rosvold et al. (1956)) is among the tasks most frequently used to study adaptive cognitive control by cognitive and clinical neuroscientists (Cohen and Servan-Schreiber,1992; Servan-Schreiber et al.,1996). In particular, the task makes it possible to distinguish between proactive or reactive control modes (Braver (2012); Braver et al. 2007).
Test of Emotion Comprehension (TEC) | Six months: Change in TEC from baseline to 6 months follow-up measured by lab assessment.
  The TEC is a direct assessment measure used to capture child emotion understanding (Kårstad et al., 2015; Pons & Harris, 2000). The TEC measures nine components of emotion understanding: 1) emotion recognition, 2) external cause, 3) desire, 4) belief, 5) reminder, 6) regulation, 7) hidden, 8) mixed, and 9) morally based emotions.

CONTACTS AND LOCATIONS:
Overall Officials: Evalill Bølstad, PhD, Principal Investigator — University of Oslo
Locations (1):
- University of Oslo, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided